CLINICAL TRIAL: NCT02015234
Title: A 12-Month, Multicenter, Open-Label Extension Study (F202) to Evaluate the Long-term Safety of TNX-102 SL Tablets Taken Daily at Bedtime in Patients With Fibromyalgia
Brief Title: 12-Month Open-Label Long-term Safety Study of TNX-102 SL Tablets in Fibromyalgia Patients
Acronym: BESTFIT-OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-F203
Record Dates: First submitted 2013-12-09; First posted 2013-12-19 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Primary Fibromyalgia
Keywords: TNX-102 SL; bedtime; sublingual; 12-month; long term safety; long term efficacy; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TNX-102 SL (Experimental): 1x TNX-102 SL 2.8 mg sublingual tablet taken daily at bedtime for 12 months
  Interventions: Drug: TNX-102 SL

INTERVENTIONS:
Drug: TNX-102 SL — TNX-102 SL 2.8 mg taken daily at bedtime.
  Other Names: cyclobenzaprine HCl

SUMMARY:
This was an open-label, extension trial designed to evaluate the long-term safety over 12 months of TNX-102 SL tablets taken daily at bedtime for the treatment of fibromyalgia. Patients recruited into this trial were those who had successfully completed the double-blind study, TNX-CY-F202 (F202) (NCT01903265). Patients were not made aware of the therapy they received during the double-blind study.

DETAILED DESCRIPTION:
The study consisted of 7 clinic visits, including Screening/Baseline Visit 1 (Day 0 which was typically the same date as Visit 6 of the double-blind lead-in study), visits after 1, 3, 6, 9, and 12 months of treatment (Visits 2-6), and a Follow-up Visit (Visit 7) scheduled within one month after stopping study drug treatment.

Primary:

The primary objective of the study was to evaluate the long-term safety of TNX-102 SL tablets taken daily at bedtime over 12 months in patients with fibromyalgia who have completed Study TNX-CY-F202 (NCT01903265)

Secondary:

The secondary objective was to evaluate the long-term efficacy of TNX-102 SL tablets taken daily at bedtime to control symptoms of fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

1. The patient met all prior inclusion and exclusion requirements for Study F202 (NCT01903265) originally, and has had no intervening medical conditions, increased suicidal ideation, or requirements for concomitant medications that preclude exposure to TNX-102 SL or enrollment in the extension study.
2. The patient completed expected dosing in F202 (NCT01903265) defined as taking study medication up to Week 12, with at least 70% compliance with medication usage (based on responses from daily IVRS calls recorded during the F202 study (NCT01903265)) and no major protocol violations.
3. The patient has provided written informed consent to participate in this extension protocol.

Exclusion Criteria:

None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, Study Director — Tonix Pharmaceuticals
Locations (13):
- United States (13):
  - Denver, Denver, Colorado
  - 16176 Cortez Boulevard, Brooksville, Florida
  - 100 West Gore Street, Orlando, Florida
  - 71 Thomas Johnson Drive, Frederick, Maryland
  - 370 Faunce Corner Road, North Dartmouth, Massachusetts
  - Worcester, Worcester, Massachusetts
  - Jackson, Jackson, Mississippi
  - Cincinnati, Cincinnati, Ohio
  - 1275 Olentangy River Road, Columbus, Ohio
  - 18660 Bagley Road, Middleburg Heights, Ohio
  - 1001 South Market Street, Mechanicsburg, Pennsylvania
  - 322 Memorial Drive, Greer, South Carolina
  - 601 Broadway, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred fifty-eight (158) of the 174 patients who completed 12 weeks of treatment in Study F202 were eligible and consented to participate in the 12-month safety extension study.
Pre-assignment Details: Restricted to patients who completed the lead-in double-blind study and continued to meet the inclusion/exclusion criteria.
Groups:
- Placebo - TNX-102 SL 2.8 mg: These patients received placebo during the lead-in study (F202), followed by 1 x TNX-102 SL 2.8 mg tablet taken daily at bedtime for 12 months during the open-label study.
- TNX-102 SL 2.8mg - TNX-102 SL 2.8 mg: These patients received 1 x TNX-102 SL 2.8 mg tablet taken daily at bedtime during both the lead-in study (F202) as well as the open-label study, for a total treatment duration of up to 15 months.
Period: Overall Study
Arm/Group | Placebo - TNX-102 SL 2.8 mg | TNX-102 SL 2.8mg - TNX-102 SL 2.8 mg
Started | 79 | 79
Completed | 43 | 54
Not Completed | 36 | 25

BASELINE CHARACTERISTICS:
Groups:
- Placebo - TNX-102 SL 2.8 mg; TNX-102 SL 2.8 mg - TNX-102 SL 2.8 mg: 1x TNX-102 SL 2.8 mg sublingual tablet taken daily at bedtime for 12 months
  TNX-102 SL: TNX-102 2.8 mg SL taken daily at bedtime.
- Total: Total of all reporting groups
Arm/Group | Placebo - TNX-102 SL 2.8 mg | TNX-102 SL 2.8 mg - TNX-102 SL 2.8 mg | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 79 | 154
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Full Range); unit: Years] | 50.2 [19 to 65] | 51.7 [20 to 64] | 50.9 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 153
  Male | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Newly-emergent Adverse Events (NEAEs) During Treatment With TNX-102 SL Tablets Taken Daily at Bedtime Over 12 Months in Patients With Fibromyalgia.
Description: NEAEs and Serious Adverse events (SAEs) were collected and are coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: Up to 12 months
Population: All of the 158 enrolled patients took at least 1 dose of study drug and were included in the safety analysis population.
Measure: Count of Participants; unit: Participants
Groups:
- TNX-102 SL 2.8 mg - TNX-102 SL 2.8 mg: These patients received 1 x TNX-102 SL 2.8 mg tablet taken daily at bedtime during both the lead-in study (F202) as well as the open-label study, for a total treatment duration of up to 15 months.
Arm/Group | Placebo - TNX-102 SL 2.8 mg | TNX-102 SL 2.8 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 79 | 79
Participants
  Patient with at least 1 NEAE reported | 60 | 54
  Patients withdrew due to NEAE | 18 | 9
  Patient with at least 1 SAE | 3 | 5

2. Secondary Outcome: Change From Baseline in Numerical Rating Scale (NRS) Assessments of Average Pain Based on 24 Hour Recall
Description: The NRS for average pain was an 11-point scale (0=no pain → 10=worst pain imaginable) that was assessed on a 24-hour recall basis.
Time Frame: Months 1, 3, 6, 9 and 12.
Population: Patients who took at least 1 dose of study drug prior to study discontinuation were included in the efficacy analysis. By the end of the study, 36 patients from the Placebo - TNX-102 SL group and 25 patients from the TNX-102 SL - TNX-102 SL group had discontinued the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- TNX-102 SL 2.8 mg - TNX-102 SL 2.8 mg: These patients received 1 x TNX-102 SL 2.8 mg tablet taken daily at bedtime during both the lead-in study (F202), as well as the open-label study, for a total treatment duration of up to 15 months.
Arm/Group | Placebo - TNX-102 SL 2.8 mg | TNX-102 SL 2.8 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 79 | 79
Scores on a scale
  Baseline | 5.6 (2.29) | 5.0 (2.52)
  Change at Month 1: number analyzed (Participants) | 65 | 75
  Change at Month 1 | -0.5 (1.96) | -0.2 (1.75)
  Change at Month 3: number analyzed (Participants) | 56 | 63
  Change at Month 3 | -0.5 (1.86) | -0.3 (1.92)
  Change at Month 6: number analyzed (Participants) | 50 | 58
  Change at Month 6 | -0.7 (2.18) | -0.2 (2.32)
  Change at Month 9: number analyzed (Participants) | 46 | 55
  Change at Month 9 | -0.6 (2.36) | 0.0 (1.91)
  Change at Month 12: number analyzed (Participants) | 43 | 54
  Change at Month 12 | 0.1 (2.08) | -0.0 (2.26)

3. Secondary Outcome: Change From Baseline in Numerical Rating Scale (NRS) Assessments of Average Pain Based on a 7 Day Recall
Description: The NRS for average pain over the past 7 days was an 11-point scale (0=no pain → 10=worst pain imaginable) that was assessed on a 7-day recall basis.
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo - TNX-102 SL 2.8 mg | TNX-102 SL 2.8 mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 79 | 79
Scores on a scale
  Baseline | 5.7 (2.09) | 4.8 (2.18)
  Change at Month 1: number analyzed (Participants) | 65 | 75
  Change at Month 1 | -0.8 (1.68) | 0.1 (1.13)
  Change at Month 3: number analyzed (Participants) | 56 | 63
  Change at Month 3 | -0.6 (1.67) | 0.1 (1.85)
  Change at Month 6: number analyzed (Participants) | 50 | 58
  Change at Month 6 | -0.7 (2.06) | 0.2 (2.11)
  Change at Month 9: number analyzed (Participants) | 46 | 55
  Change at Month 9 | -0.4 (2.33) | 0.0 (2.07)
  Change at Month 12: number analyzed (Participants) | 43 | 54
  Change at Month 12 | 0.0 (1.72) | 0.2 (1.84)

4. Secondary Outcome: Responder Analysis of Patient's Global Impression of Change (PGIC)
Description: PGIC is a fibromyalgia-specific validated instrument to gauge the patient's assessment of change in condition.The scores are categorized as provided below. A responder was defined by a score of 1 (very much improved), or 2 (much improved).
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
Time Frame: Months 1, 3, 6, 9, 12
Population: Patients who took at least 1 dose of study drug prior to study discontinuation were included in the efficacy analysis. Overall, 36 patients from the Placebo - TNX-102 SL group and 25 patients from the TNX-102 SL - TNX-102 SL group had discontinued the study early. Any missing PGIC responses were included in the "scores 3-7" for that visit.
Measure: Count of Participants; unit: Participants
Groups:
- TNX-102 SL 2.8mg - TNX-102 SL 2.8 mg: These patients received 1 x TNX-102 SL 2.8 mg tablet taken daily at bedtime during both the lead-in study (F202), as well as the open-label study, for a total treatment duration of up to 15 months.
Arm/Group | Placebo - TNX-102 SL 2.8 mg | TNX-102 SL 2.8mg - TNX-102 SL 2.8 mg
Number analyzed (Participants) | 79 | 79
Participants
  Month 1: Score 1 or 2 | 16 | 25
  Month 1: Scores 3 to 7 | 63 | 54
  Month 3: Score 1 or 2 | 23 | 29
  Month 3: Scores 3 to 7 | 56 | 50
  Month 6: Score 1 or 2 | 22 | 26
  Month 6: Scores 3 to 7 | 57 | 53
  Month 9: Score 1 or 2 | 21 | 27
  Month 9: Scores 3 to 7 | 58 | 52
  Month 12: Score 1 or 2 | 17 | 32
  Month 12: Scores 3 to 7 | 62 | 47

ADVERSE EVENTS:
Time Frame: 12 months
Description: 5% was used as the adverse event reporting cut-off
Arm/Group | Placebo - TNX-102 SL 2.8 mg | TNX-102 SL 2.8mg - TNX-102 SL 2.8 mg
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/79
Serious Adverse Events (participants affected / at risk) | 3/79 | 5/79
Other Adverse Events (participants affected / at risk) | 43/79 | 39/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - TNX-102 SL 2.8 mg (N=79) | TNX-102 SL 2.8mg - TNX-102 SL 2.8 mg (N=79)
Anxiety (Psychiatric disorders) | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Brain stem glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pubic fracture (Injury, poisoning and procedural complications) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - TNX-102 SL 2.8 mg (N=79) | TNX-102 SL 2.8mg - TNX-102 SL 2.8 mg (N=79)
Hypoaesthesia oral (Gastrointestinal disorders) | 22 | 1
Sinusitis (Infections and infestations) | 1 | 10
Fatigue (General disorders) | 3 | 8
Product taste abnormal (General disorders) | 9 | 0
Glossodynia (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 2 | 4
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Somnolence (Nervous system disorders) | 1 | 4
Paraesthesia (Nervous system disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA in place with all study investigators.